CLINICAL TRIAL: NCT00385723
Title: Omega-3 Dietary Supplementation, Immune Function, and Mood
Brief Title: Fish Oil (Omega 3), Immune Function, and Mood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Professor of Psychiatry and Psychology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0087; 2006H0054; R01AG029562 (NIH)
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Inflammation
Keywords: affect; inflammation
MeSH Terms: conditions — Inflammation | interventions — Docosahexaenoic Acids; Fish Oils; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 1.25 g/d
  Interventions: Dietary Supplement: Omega 3 (Fish Oil) Supplementation
- 2 (Experimental): 2.496 g/d
  Interventions: Dietary Supplement: Omega 3 (Fish Oil) Supplementation
- 3 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3 (Fish Oil) Supplementation — 1.25 g or 2.496 g daily for 4 months
  Arms: 1; 2
Dietary Supplement: Placebo — matching placebo capsule daily for 4 months
  Arms: 3

SUMMARY:
This study is designed to examine the effects of fish oil on immune function and mood.

DETAILED DESCRIPTION:
The beneficial effects of fish oil (or eating fish more frequently) include reductions in triglycerides, blood pressure, and heart rate, as well as increases in HDL cholesterol, the "good" type of cholesterol. In addition, certain aspects of immune function also appear to show favorable responses to fish oil supplementation, and some studies suggest that fish oil helps to improve mood and decrease depression.

This study is designed to examine how supplementation with omega-3 polyunsaturated fatty acids (key fish oil components) affects aspects of your immune response, and your mood; because some research suggests that people who eat more fish may do better during stressful times, the study will also examine how fish oil affects your immune response to stress, certain stress hormone responses, and your psychological response to stress.

For detailed information about the study, please visit our website at http://www.stressandhealth.org

ELIGIBILITY:
Recruiting men and women ages 40-88 from the Greater Columbus Ohio area. Participation involves taking capsules for 4 months and completing 6 appointments (for a total of 19.5 hours) at Ohio State.

Inclusion Criteria:

* Healthy men and women
* NOT currently taking any sort of fish oil or omega 3 supplement

Exclusion Criteria:

* Use of blood pressure medicines, cholesterol-lowering drugs, steroids, or antidepressants
* Certain lifestyle habits such as smoking or exercising vigorously for 2 or more hours a week may also exclude applicants from participating

Ages: 40 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice K. Kiecolt-Glaser, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Kiecolt-Glaser JK, Belury MA, Andridge R, Malarkey WB, Hwang BS, Glaser R. Omega-3 supplementation lowers inflammation in healthy middle-aged and older adults: a randomized controlled trial. Brain Behav Immun. 2012 Aug;26(6):988-95. doi: 10.1016/j.bbi.2012.05.011. Epub 2012 May 26. PMID 22640930
- [Result] Kiecolt-Glaser JK, Epel ES, Belury MA, Andridge R, Lin J, Glaser R, Malarkey WB, Hwang BS, Blackburn E. Omega-3 fatty acids, oxidative stress, and leukocyte telomere length: A randomized controlled trial. Brain Behav Immun. 2013 Feb;28:16-24. doi: 10.1016/j.bbi.2012.09.004. Epub 2012 Sep 23. PMID 23010452
- [Derived] Madison AA, Belury MA, Andridge R, Renna ME, Rosie Shrout M, Malarkey WB, Lin J, Epel ES, Kiecolt-Glaser JK. Omega-3 supplementation and stress reactivity of cellular aging biomarkers: an ancillary substudy of a randomized, controlled trial in midlife adults. Mol Psychiatry. 2021 Jul;26(7):3034-3042. doi: 10.1038/s41380-021-01077-2. Epub 2021 Apr 20. PMID 33875799
- [Derived] Jaremka LM, Derry HM, Bornstein R, Prakash RS, Peng J, Belury MA, Andridge RR, Malarkey WB, Kiecolt-Glaser JK. Omega-3 supplementation and loneliness-related memory problems: secondary analyses of a randomized controlled trial. Psychosom Med. 2014 Oct;76(8):650-8. doi: 10.1097/PSY.0000000000000104. PMID 25264972
- See also: Please click here to visit our website if you would like to read more about the study or apply to participate. — http://www.stressandhealth.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data collection for this double-blind placebo-controlled four month randomized clinical trial began in September, 2006 and ended in February, 2011. Ohio State University campus and community print and web-based announcements were used for recruitment.
Pre-assignment Details: We used participants' ability to follow the regimen as a criterion for study entry. Participants received a 7-day supply of placebo capsules (single blind) at the subsequent in-person screening session, and those who had taken less than 80% of the capsules a week later were dropped before randomization.
Groups:
- Placebo: Placebo : matching placebo capsule daily for 4 months
- 1.25 g/d n-3: Omega 3 (Fish Oil) Supplementation : 1.25 g daily for 4 months
- 2.5 g/d n-3: Omega 3 (Fish Oil) Supplementation : 2.496 g daily for 4 months
Period: Overall Study
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3
Started | 46 | 46 | 46
Completed | 44 | 45 | 44
Not Completed | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3 | Total
Number analyzed (Participants) | 46 | 46 | 46 | 138
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (8.6) | 51.1 (8.0) | 51.0 (6.7) | 51.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 29 | 93
  Male | 10 | 18 | 17 | 45
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33 | 39 | 37 | 109
  Black | 9 | 5 | 8 | 22
  Asian | 2 | 1 | 1 | 4
  Other | 2 | 1 | 0 | 3
Sagittal abdominal diameter [Mean (Standard Deviation); unit: cm] | 22.8 (3.2) | 23.9 (3.4) | 22.9 (2.9) | 22.8 (3.0)
CES-D [Median (Inter-Quartile Range); unit: scores on a scale] — Center for Epidemiologic Studies Depression Scale (CES-D) score The CES-D is a self-report scale designed to measure current symptoms of depression rated on a four-point likert scale.
  Scores range from 0-60, with higher scores indicating a higher frequency of depressive symptoms.
  scores on a scale | 5 [3 to 9] | 5 [2 to 11] | 6 [2 to 10] | 5 [2 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Serum ln(TNF-a)
Description: log-transformed serum Tumor Necrosis Factor-alpha (TNF-alpha)
Time Frame: Baseline & 4 months
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: pg/ml (raw TNF-a)
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3
Number analyzed (Participants) | 46 | 46 | 46
pg/ml (raw TNF-a)
  Baseline (visit 1) | 0.66 (0.25) | 0.74 (0.25) | 0.71 (0.25)
  Change, Visit 1 to 5 | 0.11 (0.030) | 0.002 (0.028) | -0.024 (0.029)
Statistical Analysis 1: Comparison: Placebo vs 1.25 g/d n-3; Comparison was made on change from baseline to 4 months; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.11, 95% CI 2-sided [-0.19 to -0.028], Standard Error of Mean 0.04 — 1.25 g/d minus placebo
Statistical Analysis 2: Comparison: Placebo vs 2.5 g/d n-3; Comparison was made on the change from baseline to 4 months; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.13, 95% CI 2-sided [-0.22 to -0.052], Standard Error of Mean 0.04 — 2.5 g/d minus placebo

2. Primary Outcome: Serum ln(IL-6)
Description: log-transformed serum Interleukin-6 (IL-6)
Time Frame: Baseline & 4 months
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: pg/ml (raw IL-6)
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3
Number analyzed (Participants) | 46 | 46 | 46
pg/ml (raw IL-6)
  Baseline (visit 1) | 0.91 (0.60) | 1.02 (0.60) | 0.85 (0.60)
  Change, Visit 1 to 5 | 0.31 (0.077) | -0.106 (0.070) | -0.123 (0.074)
Statistical Analysis 1: Comparison: Placebo vs 1.25 g/d n-3; Comparison was made on change from baseline to 4 months; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.41, 95% CI 2-sided [-0.62 to -0.21], Standard Error of Mean 0.10 — 1.25 g/d minus placebo
Statistical Analysis 2: Comparison: Placebo vs 2.5 g/d n-3; Comparison was made on the change from baseline to 4 months; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.43, 95% CI 2-sided [-0.64 to -0.22], Standard Error of Mean 0.11 — 2.5 g/d minus placebo

3. Primary Outcome: ln(CES-D)
Description: log-transformed Center for Epidemiologic Studies Depression Scale (CES-D) score The CES-D is a self-report scale designed to measure current symptoms of depression rated on a four-point likert scale.
  Scores range from 0-60, with higher scores indicating a higher frequency of depressive symptoms.
Time Frame: Baseline & 4 months
Population: intention to treat
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3
Number analyzed (Participants) | 46 | 46 | 46
scores on a scale
  Baseline (visit 1) | 1.5 (0.17) | 1.5 (0.17) | 1.6 (0.17)
  Change, visit 1 to 5 | -0.056 (0.15) | -0.29 (0.15) | -0.26 (0.15)
Statistical Analysis 1: Comparison: Placebo vs 1.25 g/d n-3; Comparison was made on the change from baseline to 4 months; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.23, 95% CI 2-sided [-0.64 to 0.18], Standard Error of Mean 0.21 — 1.25 g/d minus placebo
Statistical Analysis 2: Comparison: Placebo vs 2.5 g/d n-3; Comparison was made on the change from baseline to 4 months; Test type: Superiority or Other; p = 1.0, Mixed Models Analysis — Bonferroni-adjusted to account for multiple testing; Difference in change from baseline = -0.20, 95% CI 2-sided [-0.61 to 0.21], Standard Error of Mean 0.21 — 2.5 g/d minus placebo

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Placebo | 1.25 g/d n-3 | 2.5 g/d n-3
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 42/46 | 38/46 | 40/46
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=46) | 1.25 g/d n-3 (N=46) | 2.5 g/d n-3 (N=46)
Ear ache (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (10) | 8 (8)
Swollen glands (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 20 (20) | 23 (23)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) | 6 (6)
Wet cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 8 (8)
Stomach pain (Gastrointestinal disorders) | 12 (12) | 13 (13) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 10 (10) | 7 (7) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes